CLINICAL TRIAL: NCT01479764
Title: Effect of Sugammadex Compared With Usual Care for Reversal of Neuromuscular Blockade Induced by Rocuronium on Incidence of Residual Blockade at PACU Entry
Brief Title: Study of Sugammadex Versus Usual Care on Incidence of Residual Blockade at Post Anesthesia Care Unit Admission (P07981)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07981; MK-8616-064 (Other: Merck study number)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2013-12-31 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Surgical Procedures, Elective
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): Participants receive sugammadex, 2 or 4 mg/kg, depending on level of neuromuscular recovery
  Interventions: Drug: Sugammadex
- Neostigmine/glycopyrrolate (Active Comparator): Participants receive neostigmine/glycopyrrolate per usual practice
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Sugammadex — sugammadex, intravenous (IV) bolus, 2 or 4 mg/kg depending on level of neuromuscular recovery
  Other Names: SCH 900616, MK-8616
  Arms: Sugammadex
Drug: Neostigmine — neostigmine, per usual practice
  Arms: Neostigmine/glycopyrrolate
Drug: Glycopyrrolate — glycopyrrolate per usual practice
  Arms: Neostigmine/glycopyrrolate

SUMMARY:
This study will compare the incidence of residual neuromuscular blockade in participants who undergo reversal of neuromuscular blockade with sugammadex compared to those who undergo reversal of neuromuscular blockade with usual care (neostigmine/glycopyrrolate).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 or 2 or 3
* Scheduled to undergo an elective abdominal surgical procedure under general anesthesia; and:

  * expected to undergo neuromuscular relaxation with rocuronium for

endotracheal intubation; and

* expected to require at least one maintenance dose of rocuronium; and
* expected to require active reversal of neuromuscular blockade; and
* expected to require clinical or subjective neuromuscular monitoring only; and
* expected to recover in the PACU

  * Arm that is accessible for measuring the TOF ratio in the PACU
  * Sexually active female patient of child-bearing potential must agree to use a

medically accepted method of contraception through seven days after receiving

protocol-specified medication.

Exclusion Criteria:

* Anatomical malformations that may lead to difficult intubation
* Neuromuscular disorder(s) that may affect neuromuscular blockade and/or trial assessments
* Dialysis-dependent or has or is suspected of having severe renal insufficiency
* Significant hepatic dysfunction
* Family history of malignant hyperthermia
* Cardiac pacemaker
* Allergy to study treatments or its/their excipients, to opioids / opiates, sugammadex, muscle relaxants or their excipients, or other medication(s) used during general anesthesia
* Toremifene before or within 24 hours of study drug administration
* Scheduled for an overnight stay (or >12 hours) in PACU
* Expected transfer to an Intensive Care Unit after surgery
* Pregnant, intention to become pregnant between randomization and the Day 30 pregnancy follow-up visit
* Breast-feeding.
* Investigational drug(s) within 30 days of randomization on this study
* Participation in any other clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial
* Participant or family member is among the personnel of the investigational or Sponsor staff directly involved with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-12-02 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2012-11-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Brueckmann B, Sasaki N, Grobara P, Li MK, Woo T, de Bie J, Maktabi M, Lee J, Kwo J, Pino R, Sabouri AS, McGovern F, Staehr-Rye AK, Eikermann M. Effects of sugammadex on incidence of postoperative residual neuromuscular blockade: a randomized, controlled study. Br J Anaesth. 2015 Nov;115(5):743-51. doi: 10.1093/bja/aev104. Epub 2015 May 2. PMID 25935840

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: Participants receive a single intravenous (IV) bolus dose of sugammadex, 2 or 4 mg/kg, depending on level of neuromuscular recovery
- Neostigmine/Glycopyrrolate: Participants receive a single IV bolus dose of neostigmine/glycopyrrolate (neostigmine total dose not to exceed 5 mg) per usual practice
Period: Randomized
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Started | 76 | 78
Completed | 74 (2 randomized participants did not receive study drug) | 77 (1 randomized participant did not receive study drug)
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Treated
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Started | 74 | 77
Completed | 74 | 75
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate | Total
Number analyzed (Participants) | 74 | 77 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (12.8) | 57.0 (12.7) | 56.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Residual Neuromuscular Blockade (NMB) as Defined by a Train-of-Four (TOF) Ratio <0.9 at Post Anesthesia Care Unit (PACU) Entry
Description: Neuromuscular functioning was monitored by applying four TOF electrical stimulations to the ulnar nerve and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the magnitudes (height) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB, with a higher ratio indicating greater recovery from NMB. A T4/T1 Ratio of <0.9 is indicative of residual NMB.
Time Frame: At PACU entry on Day 1
Population: The analysis population consisted of all randomized participants who received at least one dose of study drug (sugammadex or neostigmine/glycopyrrolate) and had a reliable TOF measurement at PACU entry.
Measure: Number; unit: participants
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 74 | 76
participants | 0 | 33
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine/Glycopyrrolate; Sugammadex is the numerator and Neostigmine/Glycopyrrolate is the denominator; Test type: Superiority or Other; p < 0.0001, Pearson's Chi-square test; Odds Ratio (OR) = 0.0, 95% CI 2-sided [0.000 to 0.059]

2. Secondary Outcome: Time From Start of Study Drug Administration to Operating Room Discharge-ready
Description: The time of operating room discharge readiness was determined by the surgical team based on clinical evaluations.
Time Frame: Day 1
Population: The analysis population consisted of all randomized participants who received at least one dose of study drug (sugammadex or neostigmine/glycopyrrolate).
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 74 | 77
minutes | 15.02 [13.23 to 17.05] | 18.05 [15.94 to 20.43]
Statistical Analysis 1: Comparison: Sugammadex vs Neostigmine/Glycopyrrolate; Sugammadex is the numerator and neostigmine/glycopyrrolate is the denominator. Used log-transformed time intervals; Test type: Superiority or Other; p = 0.021, ANCOVA; Adjusted for age, American Society of Anesthesiologists class, Body Mass Index, comorbidity index & length of surgical procedure; Estimated Ratio of Geometric Means = 0.83, 95% CI 2-sided [0.71 to 0.97]

ADVERSE EVENTS:
Time Frame: Up to 7 days after administration of study drug
Description: Treatment emergent adverse events in the All Patients as Treated population which consisted of all randomized participants who received at least one dose of study drug (sugammadex or neostigmine/glycopyrrolate).
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Serious Adverse Events (participants affected / at risk) | 7/74 | 8/77
Other Adverse Events (participants affected / at risk) | 18/74 | 18/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=74) | Neostigmine/Glycopyrrolate (N=77)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastronintestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 3 (3)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=74) | Neostigmine/Glycopyrrolate (N=77)
Bradycardia (Cardiac disorders) | 0 (0) | 4 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 6 (6) | 6 (7)
Hypertension (Vascular disorders) | 10 (10) | 2 (2)
Hypotension (Vascular disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the Sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication and slides and texts of oral or other presentations that report any results of the trial.